CLINICAL TRIAL: NCT05308472
Title: (AURORA) A Randomized, Double-blind, Placebo-Controlled Study of Bitopertin to Evaluate the Safety, Tolerability, Efficacy, and Protoporphyrin IX (PPIX) Concentrations in Participants With Erythropoietic Protoporphyria (EPP)
Brief Title: Study of Bitopertin to Evaluate the Safety, Tolerability, Efficacy, and PPIX Concentrations in Participants With EPP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Disc Medicine, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: DISC-1459-201
Record Dates: First submitted 2022-03-21; First posted 2022-04-04 (Actual); Results first posted 2026-01-08 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-12

CONDITIONS: Erythropoietic Protoporphyria
Keywords: EPP; DISC-1459; RO4917838; porphyria
MeSH Terms: conditions — Protoporphyria, Erythropoietic; Porphyrias | interventions — (4-(3-fluoro-5-trifluoromethylpyridin-2-yl)piperazin-1-yl)(5-methanesulfonyl-2-(2,2,2-trifluoro-1-methylethoxy)phenyl)methanone

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- DISC-1459 oral dose level 1 (Experimental)
  Interventions: Drug: DISC-1459
- DISC-1459 oral dose level 2 (Experimental)
  Interventions: Drug: DISC-1459

INTERVENTIONS:
Drug: DISC-1459 — Oral dose level 1, once a day for 120 days
  Other Names: Bitopertin; RO4917838
  Arms: DISC-1459 oral dose level 1
Drug: DISC-1459 — Oral dose level 2, once a day for 120 days
  Other Names: Bitopertin; RO4917838
  Arms: DISC-1459 oral dose level 2
Drug: Placebo — Oral dose, once a day for 120 days
  Arms: Placebo

SUMMARY:
This is a Phase 2, multi-center, double-blind, placebo-controlled, parallel group study of bitopertin to evaluate the safety, tolerability, efficacy, and PPIX concentration change in participants with EPP. Participants may roll over to an open label extension portion after completing the double-blind treatment period.

ELIGIBILITY:
Inclusion Criteria:

1. Aged 18 years or older at the time of signing the informed consent form (ICF).
2. Diagnosis of EPP, based on medical history by ferrochelatase ( FECH) genotyping or by biochemical porphyrin analysis.
3. Body weight ≥50 kg.
4. Washout of at least 2 months prior to Screening of afamelanotide and dersimelagon, if applicable.
5. Aspartate aminotransferase (AST) and alanine transaminase (ALT) <2× upper limit of normal (ULN) and total bilirubin <ULN (unless documented Gilbert syndrome) at Screening. Albumin >lower limit of normal (LLN).

Exclusion Criteria:

Medical History:

1. Major surgery within 8 weeks before Screening or incomplete recovery from any previous surgery.
2. Other than EPP, an inherited or acquired red cell disease associated with anemia.
3. A history or known allergic reaction to any investigational product excipients or history of anaphylaxis to any food or drug.
4. History of liver transplantation.
5. History of alcohol dependence or excessive alcohol consumption, as assessed by the Investigator.
6. Human immunodeficiency virus (HIV), active Hepatitis B, or C.
7. Other medical or psychiatric condition or laboratory finding not specifically noted above that, in the judgment of the Investigator or Sponsor, would put the participant at unacceptable risk or otherwise preclude the participant from participating in the study
8. Condition or concomitant medication that would confound the ability to interpret clinical, clinical laboratory, or participant diary data, including a major psychiatric condition that has had an exacerbation or required hospitalization in the last 6 months.

   Treatment History:
9. Concurrent or planned treatment with afamelanotide or dersimelagon during the study period.
10. Treatment with opioids for any period >7 days in the 2 months prior to screening or anticipated to require opioid use for >7 days at any point during the study.
11. New treatment for anemia, including initiation of iron supplementation, in the 2 months prior to Screening.
12. Current or planned use of any drugs or herbal remedies known to be strong inhibitors or inducers of CYP3A4 enzymes for 28 days prior to the first dose and throughout the study.

    Laboratory Exclusions:
13. Hemoglobin <10 g/dL at Screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2022-10-31 (Actual); Primary Completion 2024-02-20 (Actual); Study Completion 2024-08-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Will Savage, MD PhD, Study Director — Disc Medicine
Locations (9):
- United States (9):
  - University of Alabama Hospital, Birmingham, Alabama
  - University of California San Francisco, San Francisco, California
  - University of Miami Miller School of Medicine, Miami, Florida
  - Massachusetts General Hospital, Boston, Massachusetts
  - Mount Sinai Hospital, New York, New York
  - Atrium Health Wake Forest Baptist, Winston-Salem, North Carolina
  - Einstein Medical Center, Philadelphia, Pennsylvania
  - University of Texas, Galveston, Texas
  - Fred Hutchinson Cancer Center, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- DISC-1459 Oral Low Dose: DISC-1459: Oral 20 mg, once a day for 120 days
- DISC-1459 Oral High Dose: DISC-1459: Oral 60 mg, once a day for 120 days
Period: Overall Study
Arm/Group | Placebo | DISC-1459 Oral Low Dose | DISC-1459 Oral High Dose
Started | 24 | 26 | 25
Completed | 24 | 26 | 22
Not Completed | 0 | 0 | 3
Not completed — Adverse Event | 0 | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- DISC-1459 Oral Low Dose Level: DISC-1459: Oral 20 mg dose, once a day for 120 days
- DISC-1459 Oral High Dose Level: DISC-1459: Oral 60 mg dose, once a day for 120 days
- Total: Total of all reporting groups
Arm/Group | Placebo | DISC-1459 Oral Low Dose Level | DISC-1459 Oral High Dose Level | Total
Number analyzed (Participants) | 24 | 26 | 25 | 75
Age, Customized [Mean (Standard Deviation); unit: years]
  Age | 42.3 (12.24) | 45.0 (14.31) | 47.8 (14.02) | 45.1 (13.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 14 | 12 | 38
  Male | 12 | 12 | 13 | 37
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 0 | 2 | 4
  Not Hispanic or Latino | 22 | 26 | 23 | 71
  Unknown or Not Reported | 0 | 0 | 0 | 0
Whole Blood Metal-free PPIX [Mean (Standard Deviation); unit: ng/mL] — Baseline PPIX concentrations consist of the average of all measurable concentrations prior to first dose of study drug.
  ng/mL | 8691.0 (424.56) | 8154.6 (6816.49) | 10597.0 (4916.24) | 9140.4 (5544.78)

OUTCOME MEASURES:

1. Primary Outcome: Percent Change From Baseline in Whole Blood Metal-free PPIX Levels
Description: Percent change from baseline in PPIX concentration was analyzed using a mixed model repeated measures analysis in the ITT population.
Time Frame: 121 days
Measure: Mean (95% Confidence Interval); unit: Percent Change
Groups:
- DISC-1459 Oral Low Dose: DISC-1459: Oral 20 mg dose, once a day for 120 days
- DISC-1459 Oral High Dose l: DISC-1459: Oral 60 mg dose, once a day for 120 days
Arm/Group | Placebo | DISC-1459 Oral Low Dose | DISC-1459 Oral High Dose l
Number analyzed (Participants) | 24 | 26 | 25
Percent Change | 8.07 [-6.200 to 22.338] | -21.48 [-35.842 to -7.125] | -41.74 [-56.531 to -26.950]

2. Secondary Outcome: Total Hours of Sunlight Exposure to Skin on Days With no Pain From 1000 to 1800 Hours (10:00am to 6:00pm)
Description: Cumulative total hours of sunlight exposure on days with no pain from 1000 to 1800 hours from baseline to Day 121 (EOS) was analyzed using analysis of variance in the ITT population.
Time Frame: 121 days
Measure: Mean (95% Confidence Interval); unit: Hours
Arm/Group | Placebo | DISC-1459 Oral Low Dose Level | DISC-1459 Oral High Dose Level
Number analyzed (Participants) | 24 | 26 | 25
Hours | 133.91 [92.180 to 175.643] | 175.11 [134.723 to 215.489] | 153.14 [111.699 to 194.585]

3. Secondary Outcome: Daily Sunlight Exposure Time (Minutes) to First Prodromal Symptom (Burning, Tingling, Itching, or Stinging) Associated With Sunlight Exposure Between 1 Hour Post-sunrise and 1 Hour Pre-sunset
Description: Participants exposed their skin to sunlight once a week and measured the time it takes to experience a prodrome. The time (minutes) to first prodromal symptom (e.g., burning, tingling, itching, or stinging) associated with sunlight exposure was recorded in a diary. This sun exposure challenge was performed weekly. The average time (minutes) to first prodromal symptom (e.g., burning, tingling, itching, or stinging) associated with sunlight exposure was averaged over two-week intervals through Study Day 121.
Time Frame: 121 days
Measure: Mean (Standard Deviation); unit: Minutes/Two Weeks
Groups:
- DISC-1459 Oral High Dose: DISC-1459: Oral 60 mg dose, once a day for 120 days
Arm/Group | Placebo | DISC-1459 Oral Low Dose | DISC-1459 Oral High Dose
Number analyzed (Participants) | 20 | 22 | 20
Minutes/Two Weeks | 149.05 (116.434) | 155.51 (99.903) | 176.14 (134.952)

4. Secondary Outcome: Total Pain Intensity
Description: The maximum total daily pain intensity scores of phototoxic reactions over the entire treatment period (D1-D121). The maximum pain score of a phototoxic reaction was measured on a Likert Scale (0-10). Total scores range from 0-1210. A score of "0" is the best outcome; and higher scores are a worse outcome. The maximum pain values on a scale of 0-10 in a day were summed across 121 days.
Time Frame: Sum of Day 1 to Day 121
Measure: Mean (Standard Deviation); unit: Scores on a scale
Groups:
- Placebo: Placebo: Oral dose, once a day for 121 days
- DISC-1459 Oral Low Dose Level: DISC-1459: Oral 20 mg dose, once a day for 121 days
- DISC-1459 Oral High Dose Level: DISC-1459: Oral 60 mg dose, once a day for 121 days
Arm/Group | Placebo | DISC-1459 Oral Low Dose Level | DISC-1459 Oral High Dose Level
Number analyzed (Participants) | 24 | 26 | 25
Scores on a scale | 13.0 (9.38) | 15.0 (13.95) | 6.3 (2.50)

5. Secondary Outcome: Incidence of Treatment-emergent Adverse Events
Description: Incidence of treatment-emergent adverse events
Time Frame: 121 days
Population: Number and Proportion of Participants with at Least One TEAE
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | DISC-1459 Oral Low Dose | DISC-1459 Oral High Dose
Number analyzed (Participants) | 24 | 26 | 25
Participants | 19 | 19 | 22

6. Secondary Outcome: Erythrocyte Total PPIX Concentrations
Description: Percent change from baseline in erythrocyte total PPIX concentration was summarized by analysis visit in the ITT population.
Time Frame: 121 days
Population: Intention-to-treat population analyzed
Measure: Mean (Standard Deviation); unit: Percent Change
Groups:
- DISC-1459 Oral Low Dose: DISC-1459: Oral 20 mg, once a day for 121 days
- DISC-1459 Oral High Dose: DISC-1459: Oral 60 mg, once a day for 121 days
Arm/Group | Placebo | DISC-1459 Oral Low Dose | DISC-1459 Oral High Dose
Number analyzed (Participants) | 20 | 19 | 17
Percent Change | 19.3 (59.95) | -20.5 (29.73) | -39.9 (34.67)

7. Secondary Outcome: Plasma Total PPIX Concentrations
Description: Percent change from baseline in plasma total PPIX concentration was summarized by analysis visit in the ITT population.
Time Frame: 121 days
Population: Intention-to-treat population analyzed
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo | DISC-1459 Oral Low Dose Level | DISC-1459 Oral High Dose Level
Number analyzed (Participants) | 18 | 18 | 13
Percent Change | 11.7 (56.76) | -45.4 (23.86) | -53.9 (31.55)

8. Secondary Outcome: Whole Blood Total PPIX Concentrations
Description: Percent change from baseline in whole blood total PPIX concentration was summarized by analysis visit in the ITT population.
Time Frame: 121 days
Population: Intention-to-treat population analyzed
Measure: Mean (Standard Deviation); unit: Percent Change
Arm/Group | Placebo | DISC-1459 Oral Low Dose Level | DISC-1459 Oral High Dose Level
Number analyzed (Participants) | 24 | 25 | 18
Percent Change | 8.2 (41.19) | -19.7 (31.71) | -40.1 (28.89)

9. Secondary Outcome: Plasma Bitopertin Concentrations
Description: Day 29 plasma bitopertin concentrations, 4 hours post-dose
Time Frame: Day 29
Population: Intention-to-treat population analyzed. There is no measurable bitopertin concentrations in placebo patients, since they did not receive drug.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | DISC-1459 Oral Low Dose Level | DISC-1459 Oral High Dose Level | Placebo
Number analyzed (Participants) | 26 | 25 | 0
ng/mL | 207.3 (83.5) | 683.4 (308.8) |

ADVERSE EVENTS:
Time Frame: 121 days
Arm/Group | Placebo | DISC-1459 Oral Low Dose Level | DISC-1459 Oral High Dose Level
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/26 | 0/25
Serious Adverse Events (participants affected / at risk) | 1/24 | 0/26 | 0/25
Other Adverse Events (participants affected / at risk) | 19/24 | 19/26 | 22/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=24) | DISC-1459 Oral Low Dose Level (N=26) | DISC-1459 Oral High Dose Level (N=25)
acute biliary pancreatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=24) | DISC-1459 Oral Low Dose Level (N=26) | DISC-1459 Oral High Dose Level (N=25)
Dizziness (Nervous system disorders) | 3 (3) | 4 (4) | 11 (11)
Headache (Nervous system disorders) | 3 (3) | 3 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 4 (4) | 1 (1) | 4 (4)
Alanine aminotransferase increased (Investigations) | 3 (3) | 1 (1) | 2 (2)
Diarrhoea (Gastrointestinal disorders) | 2 (2) | 1 (1) | 1 (1)
COVID-19 (Infections and infestations) | 2 (2) | 2 (2) | 1 (1)
Aspartate aminotransferase increased (Investigations) | 1 (1) | 1 (1) | 2 (2)
Blood iron increased (Investigations) | 0 (0) | 2 (2) | 3 (3)
Transferrin saturation increased (Investigations) | 0 (0) | 2 (2) | 2 (2)
Fatigue (General disorders) | 3 (3) | 2 (2) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-08-11): https://cdn.clinicaltrials.gov/large-docs/72/NCT05308472/Prot_SAP_002.pdf